CLINICAL TRIAL: NCT02455544
Title: The Clinical Utility of the Congo-Red Dot Test for Diagnosis and Early Prediction of Preeclampsia During Pregnancy
Status: Completed | Type: Observational
Sponsor: Catalin S Buhimschi, MD (Other)
Responsible Party: Sponsor-Investigator, Catalin S Buhimschi, MD, Director, Division of Maternal Fetal Medicine Vice-Chair, Department of Obstetrics and Gynecology, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: CRD002
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Preeclampsia
Keywords: Urine congophilia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples With DNA — Urine specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant Women: Any pregnant women that is referred to or presents to our tertiary care facility with concern for preeclampsia, will have a Congo Red Dot test preformed by research nurses. The research nurses are not involved in patient management and the results are blinded to the clinical providers and have no impact on clinical diagnosis or patient management.

SUMMARY:
The aim of the study is to validate in a prospective fashion the value of the Congo-Red Dot (CRD) test for diagnosis of preeclampsia. The working hypothesis is that in pregnancies complicated by preeclampsia, will display urine congophilia and have a positive CRD test.

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-specific hypertensive disorder and a leading cause of maternal and perinatal morbidity and death worldwide. When left untreated, preeclampsia leads to seizures (eclampsia), stroke, hemorrhage, kidney and liver failure, and death. The World Health Organization (WHO) estimates that 99% of preeclampsia-related deaths occur in low- and mid-income countries. Although most cases of maternal death are preventable, it is estimated that ~63,000 women die annually due to preeclampsia alone.

In developed countries, such as the U.S. and UK, development and implementation of clinical guidelines for diagnosis and management of preeclampsia has resulted in a dramatic decrease in maternal morbidity and mortality. Some of these measures include: a) blood pressure and dipstick proteinuria screening during each prenatal visits; b) extensive laboratory work-up to rule-out hemolysis, elevated liver enzymes, and thrombocytopenia (HELLP) syndrome; c) hospital admission for intensive clinical observation; d) use of magnesium sulfate and anti-hypertensive medication to prevent eclampsia and intracranial hemorrhage and e) medically indicated early delivery for strict clinical criteria of severity given that delivery is the only definitive cure for preeclampsia.

It is well-recognized that the number of medically-indicated early deliveries in the U.S. and U.K. exceeds those necessary to prevent maternal death or morbidity related to preeclampsia. However, in the era of widespread use of antenatal corticosteroids and advances in neonatal intensive care, in developed countries, obstetricians lean more towards indicating delivery than they were three decades ago. At present in the U.S., preeclampsia is estimated to trigger 70% of medically indicated preterm births. Yet, implementation of the same guidelines is not feasible for low- or mid-income countries. In this scenario, the tendency is to prolong pregnancy at least until 34 weeks so that the likelihood of survival for the premature neonate is maximized. Recognizing this conundrum, increased emphasis has been placed on finding novel diagnostic and prognostic biomarkers that may help with identification of preeclamptic women in real need of medically-indicated deliveries as opposed to those whose pregnancy could be safely extended. That said, for low- and mid-income countries, such biomarkers have the potential to significantly help with current barriers in reducing maternal morbidity and deaths from severe preeclampsia. Because compliance with physician referral and transport to the hospital are significant issues in rural areas, the earlier the problem is identified, the better the outcome. Accurate identification of women whose pregnancies are at high risk for preeclampsia or eclampsia would result in timely referral to medical facilities where appropriate treatments (i.e magnesium sulfate or medically-indicated delivery) can be provided. Additionally, an accurate diagnostic test for preeclampsia implemented in a developing country will allow maternity units to run more cost effectively by avoiding unnecessary referrals, unnecessary admissions for 24h protein assessment. This will also reduce the number of admissions for labor induction, the number of inductions in general and indirectly the number of C-sections.

Traditionally, the diagnosis of preeclampsia relies on presence of hypertension and proteinuria. Unfortunately, these signs are often non-specific and could be confounded by many co-morbidities including essential hypertension and chronic kidney disease. Spearheaded by proteomics research, our group identified that women with severe forms of preeclampsia excrete in their urine high amounts of unfolded or misfolded proteins. This phenomenon classifies preeclampsia as a protein conformational disorder similar to Alzheimer's and prion disease, yet particular to pregnancy. It logically followed that misfolded proteins in preeclampsia urine should exhibit congophilia (affinity for the azo-dye Congo Red). Congo Red was developed for textile industry in the 1800', but later found to have self-assembling properties and to selectively stain misfolded amyloid in brains of patients with Alzheimer's. Based on these premises, a simple urine diagnostic test [Congo Red Dot (CRD) Test] has been designed, developed and validated in our research laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women evaluated for the onset of clinical symptoms of preeclampsia in the Labor and Delivery Unit of The Ohio State Wexner Medical Center.

Exclusion Criteria:

* Non-english speaking
* Men
* Prisoners
* Those unable to provide consent for themselves

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study involves testing of urine specimens that originate from pregnant women (ages 18-48) who are presenting for evaluation, following onset of clinical symptoms of preeclampsia. Preeclampsia is a pregnancy specific medical complication of pregnancy and thus selection of specimens only of pregnant women is necessary. The urine specimens from symptomatic women will be used for the testing of the diagnosis value of the CRD test.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2014-08; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Clinical diagnosis of preeclampsia | 20 weeks gestation until 6 weeks postpartum
  Diagnostic utility of the test based on AUC

CONTACTS AND LOCATIONS:
Overall Officials: Catalin S Buhimschi, MD, Principal Investigator — The Ohio State University Department of Obstetrics and Gynecology; Irina A Buhimschi, MD, Study Director — Nationwide Children's Hospital, Center for Perinatal Research
Locations (1):
- The Ohio State Medical Center Labor and Delivery Unit, Columbus, Ohio, United States

REFERENCES:
- [Background] Buhimschi IA, Zhao G, Funai EF, Harris N, Sasson IE, Bernstein IM, Saade GR, Buhimschi CS. Proteomic profiling of urine identifies specific fragments of SERPINA1 and albumin as biomarkers of preeclampsia. Am J Obstet Gynecol. 2008 Nov;199(5):551.e1-16. doi: 10.1016/j.ajog.2008.07.006. PMID 18984079
- [Background] Buhimschi IA, Nayeri UA, Zhao G, Shook LL, Pensalfini A, Funai EF, Bernstein IM, Glabe CG, Buhimschi CS. Protein misfolding, congophilia, oligomerization, and defective amyloid processing in preeclampsia. Sci Transl Med. 2014 Jul 16;6(245):245ra92. doi: 10.1126/scitranslmed.3008808. PMID 25031267
- [Background] Buhimschi IA, Funai EF, et al. Assessment of global protein misfolding load by urine "Congo Red Dot" test for diagnosis and prediction of outcome in women with preeclampsia. Am J Obstet Gynecol 2009; 201(6A): S12.
- [Background] Buhimschi CS, Norwitz ER, Funai E, Richman S, Guller S, Lockwood CJ, Buhimschi IA. Urinary angiogenic factors cluster hypertensive disorders and identify women with severe preeclampsia. Am J Obstet Gynecol. 2005 Mar;192(3):734-41. doi: 10.1016/j.ajog.2004.12.052. PMID 15746665
- [Background] ACOG Committee on Practice Bulletins--Obstetrics. ACOG practice bulletin. Diagnosis and management of preeclampsia and eclampsia. Number 33, January 2002. Obstet Gynecol. 2002 Jan;99(1):159-67. doi: 10.1016/s0029-7844(01)01747-1. PMID 16175681